CLINICAL TRIAL: NCT07265414
Title: DRG Mutations in Prostate Cancer: a Guiding Light for Enhanced Screening and Personalised Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Fondazione Humanitas per la Ricerca (Other)
Responsible Party: Sponsor
Other Study IDs: IG 2020 ID 25027
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Bladder Cancer
Keywords: Prostate Bladder Screening DNA
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Exome analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with prostate cancer: Patients with BRCA2 variants
  Interventions: Diagnostic Test: Screening Platform

INTERVENTIONS:
Diagnostic Test: Screening Platform — Screening

SUMMARY:
At the present moment, there is no international consensus on the optimal screening to perform in men with a specific genetic/molecular risk for PCa. The number of studies exploring screening strategies tailored to men with a family history for PCa is limited [15-17]: most of them support the use of targeted screening but methodological differences make it impossible to draw conclusions from these data [18-25]. On the basis of these considerations, we believe extremely important to investigate a new approach to sort out men who will most benefit from early diagnosis. The optimization of such an approach could generate several benefits to the health service, by both reducing overdiagnosis and overtreatment in low-risk patients and decreasing the risk of underdiagnosis and undertreatment in genetically selected high-risk patients. Indeed, men with DRG mutations have higher grade and higher stage at time of diagnosis, limiting the possibility of care [2]. In the present study, we will test the hypothesis that a dedicated screening in patients with a DRG mutation, by the combination of PHI and mp-MRI, could be more effective in the PCa early detection than the current approach (DRE and PSA). We hypothesise that this targeted screening could improve the rate of early detection in PCa-positive men and increase the consequent number of curable diseases.

DETAILED DESCRIPTION:
Prostate cancer (PCa) represents the most commonly diagnosed cancer in men and the second most common cause of cancer death in Western countries. It is estimated that 5-10% of PCa cases correlate with an inherited susceptibility to the disease. Mutations in DNA-repair genes (DRGs) were found in approximately 5% of localized PCa and in 12% of metastatic castration-resistant PCa. There is an unmet clinical need to identify high risk population and distinguish truly indolent localized cancers from progressive and potentially lethal disease, which will most benefit from early diagnosis and targeted therapies, in order to avoid underdiagnosis and undertreatment in such patients. We will test whether a dedicated screening in carriers of a DRG mutation can be more effective in early detection of aggressive PCa than the current approach (PSA), increasing the number of curable diseases.

Participants will be selected according to two strategies: 1) male consanguineous relatives of women with BRCA1/2+ and/or DRG+ cancer, 2) male consanguineous relatives of men with PCa positive for a mutation in a DRG. Strategy 1 will take advantage of the large cohort of breast/ovarian cancer patients referring to our Center. Strategy 2 will involve the mutational screening by targeted NGS of DRGs on biopsy/surgical specimens with histologically-confirmed PCa and Bladder cancer (BC).

This is a monocentric, prospective study, designed to evaluate the sensitivity of a targeted screening in men at higher genetic risk for PCa because carriers of pathogenic mutations in a DNA repair gene. The study will be entirely conducted at the Istituto Clinico Humanitas throughout the collaboration of the Oncology, Urology, Pathology, Radiology Departments with the Laboratory of Medical Genetics and RNA Biology of Humanitas University

Study participants will be genetically screened for the DRG mutation they are likely to have and positive individuals will be monitored by digital rectal examination (DRE) and checking Prostate Health Index (PHI). Patients with positive DRE will receive a prostate biopsy, the others will be tested for PHI. In case of PHI>40, patients will receive an mpMRI, according to EAU guideline, and a systematic prostate biopsy plus a software fusion-guided target biopsy if mpMRI showed at least a PIRADS>2 lesion. In case of PHI 20-40, patients will undergo mpMRI and fusion-guided target biopsy when PIRADS>2 plus systematic random biopsy. Patients with a negative mpMRI (PIRADS<3) will be screened by PHI/DRE annually. In case of PHI<20, patients will be screened by DRE/PHI annually. In case of biopsy positive for PCa, patients will be consulted for precision therapy. Correlation of pathological data and clinical outcome with molecular characteristics in patients identified by our enhanced screening and in those selected by NGS analysis (i.e. positive for a DRG mutation). The latter will be follow-up as benchmark for understanding the clinical course of PCa with DRG defects

1. Select a cohort of "healthy" men with a DRG mutation and enroll them in a target screening program for early PCa detection.
2. Demonstrate that the identification of high-risk individuals can: i) detect undiagnosed PCas, ii) improve early diagnosis, iii) impact on clinical management (PARP inhibitors, immunotherapy).
3. Better understand the molecular and clinical characteristics of PCa associated with DRG defects

   * Determine the clinically significant percentage of PCa in total prostatic neoplasms;
   * Compliance to attend the "enhanced" screening (Descriptive analysis);
   * Stratification according to age at diagnosis of PCa (Descriptive analysis);
   * Correlation with pathological outcome in patients who will undergo to radical prostatectomy (Descriptive analysis + comparative analysis: ANOVA):
   * Incidence of biochemical recurrence (BCR) (Descriptive analysis)
   * Correlation of pathological data and clinical outcome (BCR) with molecular characteristics in both patients identified by our enhanced screening and those identified by the NGS analysis (i.e. positive for a DRG mutation) (Descriptive analysis + KM curves recurrence fre-survival or progression to Metastasis free survival)
   * Comparison of the mutational burden in DRG mutation positive vs. DRG mutation negative PCa (Descriptive analysis).

The responsible investigator will ensure that this study is conducted in agreement with either the Declaration of Helsinki (Tokyo, Venice, Hong Kong and Somerset West amendments) or the laws and regulations of the country, whichever provides the greatest protection of the patient. The protocol has been written, and the study will be conducted according to the ICH Guideline for Good Clinical Practice. The protocol and its annexes are subject to review and approval by the competent Independent Ethics Committee(s) ("IEC") We expect that our screening strategy will increase the rate of early diagnosis of aggressive PCa in high-risk patients and will provide useful information for targeted therapy..

ELIGIBILITY:
Inclusion Criteria:

- The following men will be screened for DRG mutations.

1. Males between the ages of 35 and 75 suffering from prostate cancer diagnosis with GS (Gleason Score) ≥ 4+3 willing to undergo screening for a mutation in one of the DNA repair genes (DRG);
2. Males under the age of 50 suffering from prostate cancer diagnosis with GS ≥ 3 +3 willing to undergo screening for a DRG mutation;
3. Consanguineous of males who, as a result of prostate biopsy and/or radical prostatectomy, have been diagnosed with prostate cancer with GS ≥ 4 + 3 and positive for a DRG mutation;
4. Consanguineous of males who following a prostate biopsy and/or radical prostatectomy had a diagnosis of prostatic cancer before the age of 50 with GS ≥ 3 +3 and positive for a DRG mutation.
5. Males and females older 18 yrs presenting with primary or secondary BC willing to undergo screening for a mutation in one of the DNA repair genes (DRG);
6. Males consanguineous of males and females who had a diagnosis of bladder cancer and positive for a DRG mutation
7. Males between the ages of 35 and 75 belonging to a family where a BRCA1/2 and/or DRG mutations has already been detected in at least one female (this screening has been and will be performed according to the AIOM 2019/NCCN 2019 guidelines, as for good clinical practice in our oncology center)

Exclusion Criteria:

-

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with relatives affected by prostate cancer
Study Population: * Contraindication absolute or relative to mpMRI
  * Active perineal/pelvic inflammatory disease
  * Urethral stricture or previous surgery for urethral surgery.
  * Subjects with chronic renal failure, marked blood protein alterations (plasma normal range 6-8 g/100 mL), hemophiliacs, or those previously submitted to multiple blood transfusions were not included in the study, as these conditions may alter the PHI analysis.
  * Any other condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Detection of prostate cancer | 5 years
  Detection of prostate cancer and screening

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Humanitas Research Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Italian Law requires a specific authorization